CLINICAL TRIAL: NCT00423033
Title: Qualitative Analysis on the Experiences of Employment Among Schizophrenic Patients
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Other Study IDs: FEMH-95-c-046
Record Dates: First submitted 2007-01-14; First posted 2007-01-17 (Estimated); Last update posted 2008-12-29 (Estimated); Status verified 2008-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The aim of this search is to realize the subjective experiences of employment among schizophrenic patients by qualitative analysis. We plan to recruit 50 people diagnosed with schizophrenia and divide into two groups, employment and unemployment. Every subjects will complete the demographic data, the evaluation of severity of disease, the record of medication and an intensive interview about their employment experiences. Finally, we will analysis the thick descriptions to understand how schizophrenic patients interpret their employment experiences and which factors will affect their successful employment.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia
* > high school

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-yen Wu, Master, Study Chair — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan